CLINICAL TRIAL: NCT02434185
Title: The Bilateral Deficit Phenomenon, Functional and Dynamometric Assessment in Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Juan Diego Ruiz-Cárdenas, BSc, MSc, Universidad Católica San Antonio de Murcia
Other Study IDs: UCAM-BLD-1
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Postmenopausal Syndrome; Muscle Weakness
Keywords: Musculoskeletal Physiological Phenomena; Postmenopause; Muscle Strength; Absorptiometry, Photon
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The bilateral deficit phenomenon (BLD) is defined as an inability of the neuromuscular system to generate maximal force when two homonymous limb operate simultaneously (bilateral contraction) with respect to the force developed when both limbs acts separately (unilateral contraction). From an applied perspective, movement patterns of bilateral homonymous limb are often developed during activities of day living, e.g. rising from a chair or opening a jar. The BLD can be considered an intrinsic property of the human neuromuscular system but could be enough important to constitute a performance-limiting factor for postmenopausal women that involves a degenerative loss of muscular strength. Therefore, a specific analysis of this phenomenon and its relation with activities of daily living, such as climbing a step and rising from a chair, is crucial for detecting variables of neuromuscular performance and develop strategies to minimize the loss of strength.

DETAILED DESCRIPTION:
* 20 postmenopausal women unexperience in strength training or resistance training, without musculoskeletal, neurological diseases, and cardiovascular limiting-diseases were recruited.
* Maximum strength of lower limbs during leg-press exercise was measured for future analysis.
* The force-time curves were measured during climbing a step and rising from a chair.
* A fragility phenotype test was applied to the subjects to determine frailty phenotype classification, including; weight loss of greater than 10 lbs in the past 12 months, maximal handgrip strength, time to walk 15-ft at usual pace, self-reported leisure time physical activity, and self-reported exhaustion.
* The anthropometric measurements were performed by dual energy X-ray absorptiometry.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women

Exclusion Criteria:

* Unexperienced in strength training or resistance training.
* Not musculoskeletal diseases.
* Not neurological diseases.
* Not cardiovascular limiting-diseases.
* Not fragility or pre-fragility phenotype.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women not experienced in strength training or resistance, without musculoskeletal, neurological diseases, and cardiovascular limiting-factor.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Assess the maximum force of lower limbs during bilateral and unilateral contraction | Screening visit
Assess the force-time curve during climbing a step | Screening visit
Assess the force-time curve during climbing rising from a chair | Screening visit
Assess bone mineral-free lean tissue mass by dual energy X-ray absorptiometry | Screening visit
Assess the fragility phenotype of the subjects | Screening visit
Assess the rate of force developed in time intervals (0-50, 50-100, 100-150ms) of lower limbs during bilateral and unilateral contraction | Screening visit
Assess fat-tissue mass and lean-tissue mass composition | Screening visit

CONTACTS AND LOCATIONS:
Overall Officials: Juan Diego JD Ruiz-Cárdenas, BSc, MSc, Principal Investigator — Universidad Católica San Antonio de Murcia
Locations (1):
- Catholic University of Murcia, Murcia, Spain

REFERENCES:
- [Derived] Ruiz-Cardenas JD, Rodriguez-Juan JJ, Jakobi JM, Rios-Diaz J, Marin-Cascales E, Rubio-Arias JA. Bilateral deficit in explosive force related to sit-to-stand performance in older postmenopausal women. Arch Gerontol Geriatr. 2018 Jan;74:145-149. doi: 10.1016/j.archger.2017.10.023. Epub 2017 Oct 31. PMID 29102831